CLINICAL TRIAL: NCT05912985
Title: Comparison of Three Different Oxygenation Strategies Consisting of Nasal Cannula, Modified Nasopharyngeal Cannula and HFNO (High Flow Nasal Oxygen) in Bronchoscopy Procedures Under Sedation
Brief Title: Three Different Oxygenation Strategies in Bronchoscopy Procedures Under Sedation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Süleyman Taş, Principal investigator, Ankara City Hospital Bilkent
Other Study IDs: SuleymanTas1
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- nasal cannula group: Nasal cannula will be used in bronchoscopy procedures in which sedation is applied in this group.
  Interventions: Other: different oxygenation methods
- modified nasopharyngeal cannula group: In this group, modified nasopharyngeal cannula will be used in bronchoscopy procedures with sedation.
  Interventions: Other: different oxygenation methods
- HFNO group: HFNO will be used in bronchoscopy procedures in which sedation is applied in this group.
  Interventions: Other: different oxygenation methods

INTERVENTIONS:
Other: different oxygenation methods — Different oxygenation methods are used in bronchoscopy procedures under sedation.

SUMMARY:
The purpose of study aims to determine which of the three different oxygenation strategies, including nasal cannula, modified nasopharyngeal cannula, and HFNO groups, is safer in patients undergoing bronchoscopy under sedation.

DETAILED DESCRIPTION:
The patients will be evaluated in the anesthesia polyclinic before the procedure, routine preparation will be made, and written informed consent will be obtained. After being informed about the study and potential risks, all patients who gave written informed consent will be enrolled in the study by recording their demographic information after determining whether they are eligible to participate in the study. In addition, STOP-BANG and FRAIL fragility questionnaires will be administered to the patients. Which oxygenation method should be used which patient will be left to the decision of the Anesthesiologist; The oxygenation tools used in the bronchoscopy unit are nasal cannula, modified nasopharyngeal cannula, and HFNO. When the patients are taken to the procedure room, anesthesia management will be applied by the standard working order of the anesthesia clinic. In addition to non-invasive arterial blood pressure monitoring, 5-channel ECG and pulse oximetry, and standard hemodynamic monitoring, Bispectral Index (BIS) monitoring will be performed. During the process, oxygen saturation will be continuously monitored and the lowest value will be recorded. Interventions made in cases of low oxygen saturation will also be recorded. At the end of the procedure, the patient will be taken to the recovery unit after waking up.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing bronchoscopy

Exclusion Criteria:

* Do not have the ability to read, understand and sign the consent form
* Pregnancy
* Contraindications to anesthetic drugs
* Hemodynamically unstable patients
* Having a peripheral vascular disease
* Intubated patients
* Patients with tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the bronchoscopy unit for the procedure
Sampling Method: Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
desaturation rate during processing | during the procedure, an average of 1 hour
  desaturation: oxygen saturation falling below 90%. Oxygen saturation was monitored continuously with a pulse oximeter attached to one of the fingers. It was recorded when oxygen saturation dropped to < 90%.

SECONDARY OUTCOMES:
rate of use of the jaw thrust maneuver during the procedure | during the procedure, an average of 1 hour
  The chin thrust maneuver is one of the maneuvers used to provide airway patency. The jaw thrust maneuvers performed by the anesthesiologist were recorded in patients who were desaturated during the procedure.
rate of airway usage during the process | during the procedure, an average of 1 hour
  The airway that was desaturated during the procedure and used by the anesthesiologist to ensure airway patency was recorded.

OTHER OUTCOMES:
Desaturation rate in patients with a high risk of Osas according to the stop-bang score | before the procedure, 2 minutes
  The stop-bang test can be used as a screening test for an osas. Scoring from 0 to 8 is given. 0-1-2 is low risk, 3-4 is medium risk, and 5-6-7-8 is high risk for Osas.
Desaturation rate in patients with higher frailty scores than frail fragility scores | before the procedure, 2 minutes
  The frail fragility test is one of the tests that measure the fragility of patients. Scoring from 0 to 5 is given. 0 is not frail, it is expressed as 1-2 prefrail and 3-4-5 frail.

CONTACTS AND LOCATIONS:
Overall Officials: süleyman taş, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No